CLINICAL TRIAL: NCT04337086
Title: The Effect of T4K Versus Twin Block in Developing Class II Division I Malocculsion (Randomized Controlled Clinical Trial)
Brief Title: Effect of T4K Versus Twin Block in Developing Class II Division I Malocculsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Dental Public Health clinical instructor and statistician, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T4k versus Twin block
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Orthodontic Appliances

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study was a double-blind study, as the participant and the outcome assessors were blinded to the type of treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T4k (Experimental)
  Interventions: Device: T4k Appliance
- Twin block (Active Comparator)
  Interventions: Device: Twin block appliance

INTERVENTIONS:
Device: T4k Appliance — The pre-fabricated, hard, polyurethane, pink T4K™ (Myo functional research Co., Australia) was used in the study. It consisted of: facial bows, lingual bows / tongue guard, lingual tag / tongue tag, dental channels with a pre-determined bite position and a lip bumper. In the first week, the patients were instructed to gradually increase the wearing time of the appliance during the daytime. By the second week, the patients were instructed to wear the appliance achieving at least 8 hours during sleeping. The Trainer usually needs no adjustments. The patients were asked to place it themselves inside their mouths. The distal ends of the appliance were trimmed 2-3 mm with an acrylic bur on a straight hand piece if they were too long or the patient could not keep his lips together. By the end of the first 4 weeks, the patients were wearing the appliances minimum of 1 hour during the day plus the overnight wear following the manufacturer's instructions.
  Arms: T4k
Device: Twin block appliance — The twin block was used, and instructions were given to wear the appliance nearly full-time. Selective sequential inter-occlusal trimming was done monthly after the 2nd month in the occlusal surface of the maxillary bite blocks to clear over the mandibular molars allowing their eruption in a more favourable mesial direction and to increase the vertical dimension. Trimming was done in the fitting surface over the maxillary and mandibular premolars whenever needed to allow their full eruption and to level the occlusal plane
  Arms: Twin block

SUMMARY:
The aim of this study was to evaluate and compare the effect of myofunctional trainer T4K versus twin block functional appliance on the dentoalveolar changes in children with class II division I malocclusion

DETAILED DESCRIPTION:
This study was a parallel arm randomized comparative clinical trial including 20 healthy children age ranged from 9-12 years showing Angle's class II division I malocclusion due to mandibular retrusion. Preoperative photographs, radiographs and study casts were taken, children were randomly assigned into two groups according to the appliance used; Group 1: T4k, and Group II: twin block. Follow up was done every 4 weeks for 9 months. Postoperative cephalometric X ray, study casts and photographs were retaken for measurements and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Angle's class II division I malocclusion due to mandibular retrusion depending on clinical judgement and confirmed with the lateral cephalometric X-ray.
* Parental written consent was secured.

Exclusion Criteria:

* Patients with mandibular shifts.
* Patients with severe crowding.
* Patients with anterior open bite.
* Patients with posterior crossbite.
* Patients with any peri-oral habits.
* Patients who had received any previous orthodontic or orthopaedic treatments.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2008-01-23 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-12-18 (Actual)

PRIMARY OUTCOMES:
Dento-alveolar changes | baseline
  This was assessed using lateral cephalometric xrays. Inclination of of maxillary incisor was assessed by measuring the angle to Frankfurt horizontal plane
Dento-alveolar changes | 9 months
  This was assessed using lateral cephalometric xrays. Inclination of of maxillary incisor was assessed by measuring the angle to Frankfurt horizontal plane
Overjet | baseline
  the extent of horizontal (anterior-posterior) overlap of the maxillary central incisors over the mandibular central incisors was measured on study casts.
Overjet | 9 months
  the extent of horizontal (anterior-posterior) overlap of the maxillary central incisors over the mandibular central incisors was measured on study casts.
Overbite | baseline
  the extent of vertical (superior-inferior) overlap of the maxillary central incisors over the mandibular central incisors, measured relative to the incisal ridges. This was assessed on study casts
Overbite | 9 months
  the extent of vertical (superior-inferior) overlap of the maxillary central incisors over the mandibular central incisors, measured relative to the incisal ridges. This was assessed on study casts

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine El Hamouly, PhD, Principal Investigator — Faculty of Dentistry, Pharos University in Alexandria.; Hanan A Ismaiel, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Azza A ElHousseiny, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Laila M El Habashy, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt